CLINICAL TRIAL: NCT04448769
Title: Epidemiological Study of Seroprevalence Against the SARS-CoV-2 Virus (COVID-19) in the Population of the Grand Nancy Metropolitan Area
Brief Title: Epidemiological Study of Seroprevalence Against the SARS-CoV-2 Virus (COVID-19)
Acronym: COVAL-NANCY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Lorraine (Other); Métropole du Grand Nancy (Unknown)
Responsible Party: Principal Investigator, Evelyne Schvoerer, Pr, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020PI128
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Coronavirus Infection; Prevalence
Keywords: Epidemiology; General population
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: A study of seroprevalence and symptom collection, or absence of symptoms, on a cluster (household) sample of the Grand Nancy Metropolitan population randomly selected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-SARS-CoV-2 IgT seropositivity (Other): Analysis of the serology result: The ELISA method allows semi-quantitative detection of total IgT antibodies. A positive sample will be defined by a ratio ≥ 1.0.
  Interventions: Biological: Anti-SARS-CoV-2 IgT seropositivity

INTERVENTIONS:
Biological: Anti-SARS-CoV-2 IgT seropositivity — Each inhabitant who agrees to participate will have to :
  * sign the consent form after receiving complete information
  * complete a questionnaire exploring sociodemographic (gender, age, professional activity...), medical (anthropometric measures, health problems, smoking...), potential contacts with COVID-19 and symptoms.
  * take a blood sample for the dermination of anti-SARS-CoV-2 IgT seropositivity of the individuals tested in the population of the Grand Nancy Metropolitan area (GNM).

SUMMARY:
In order to inform the public decision on the containment strategy and knowledge of the intensity of the epidemic during post-containment, estimates of the share of the population infected with the SARS-CoV-2 virus responsible for COVID-19 disease at the territorial level are needed as soon as possible. The aim of the study is to estimate the prevalence of positive anti-SARS-CoV-2 serologies by detection of IgT-total antibodies (IgM/IgA/IgG) in the general population of the Grand Nancy Metropolitan area.

A study of seroprevalence and symptom collection, or absence of symptoms, on a cluster (household) sample of the Grand Nancy Metropolitan population randomly selected will be conducted.

The target population consists of all the inhabitants of the Grand Nancy Metropolitan area, from which a sample is drawn from the electoral lists (households) in a random manner to ensure representativeness. In order to ultimately include 2000 people in the study

DETAILED DESCRIPTION:
In order to inform the public decision on the containment strategy and knowledge of the intensity of the epidemic during post-containment, estimates of the share of the population infected with the SARS-CoV-2 virus responsible for COVID-19 disease at the territorial level are needed as soon as possible. To date, these estimates are based on RT-qPCR tests carried out on individuals with symptoms of the disease, on people likely to present severe forms of COVID-19, known as 'vulnerable', or on the number of hospitalizations/deaths related to COVID-19. In order to refine these estimates, it is crucial to carry out measurements on a random sample of the population and to take biological samples for serological testing, in accordance with the recommendations of the HAS and the scientific societies.

Besides, it is important to assess the proportion of persons reporting that they have not developed symptoms of COVID-19 since the beginning of the epidemic among seropositive persons.

The aim of the study is to estimate the prevalence of positive anti-SARS-CoV-2 serologies by detection of IgT-total antibodies (IgM/IgA/IgG) in the general population of the Grand Nancy Metropolitan area.

A study of seroprevalence and symptom collection, or absence of symptoms, on a cluster (household) sample of the GNM population randomly selected.

It is a cross-sectional, not experimental study in the sense that it does not alter the exposure of participants; however, it does require a blood sample, which classifies it as minimal risk intervention research according to French law. The study is monocentric.

The target population consists of all the inhabitants of the Grand Nancy Metropolitan area, from which a sample is drawn from the electoral lists (households) in a random manner to ensure representativeness. In order to ultimately include 2000 people in the study.

Each inhabitant who agrees to participate will have to :

* sign the consent form after receiving complete information
* complete a questionnaire exploring sociodemographic (gender, age, professional activity...), medical (anthropometric measures, health problems, smoking...), potential contacts with COVID-19 and symptoms.
* take a blood sample:

  * in one of the identified locations of the GNM after making an appointment with the dedicated secretariat.
  * at their homes for those vulnerable to Covid-19. The total duration of participation of a subject will be ½ day (collection of consent + filling in the questionnaire and blood sampling)

Data are collected from :

* the electoral lists: surname, first names, gender, address allowing identification of the IRIS zone
* self-report questionnaires (adapted to the age : an adult questionnaire, a child questionnaire completed by the parents and an adolescent questionnaire) : socio-demographic characteristics of the respondent : age, sex, professional activity, socio-professional category, level of education ; EPICES questionnaire (adult), FAS questionnaire (child) ; medical characteristics of the respondent : weight, height, smoking status, influenza vaccination, health problems, pregnancy; potential contacts with COVID-19: perception of having been infected by the coronavirus, close relatives having been infected; potential symptoms: exploration of symptoms felt since mid-February.
* serological test results: Anti-SARS-CoV-2 IgT seropositivity

The statistical analysis concerns all participants who respond to the questionnaire (even if blood sample could not be collected); it does not include any intermediate results and there is no statistical criterion for stopping the research.

The following analyses will be carried out :

* Proportions: All proportions (including seroprevalence) will have confidence intervals calculated with the approximation by the normal distribution when the observed proportion and the size of the study group allow it, otherwise by the exact calculation of the binomial distribution.
* Risk groups: Standardized prevalences for age and sex and their confidence intervals will be given for each group of each risk factor (smoking status, weight status, level of insecurity). Significance (p-value) will be calculated by a chi-square test if the size of the subgroups allows it, a Fisher test otherwise. A relationship will be significant if p<0.05
* Analysis of the serology result: The ELISA method allows semi-quantitative detection of total IgT antibodies. A positive sample will be defined by a ratio ≥ 1.0.
* Intra-household transmission: The share of infections due to intra-household transmission will be estimated using a Bayesian model.

  * - Symptom expression groups: In seropositive participants, an exploratory study will be conducted to determine whether there are typologies of symptom expression .

This type of survey should make it possible to estimate the penetration of the virus in a very geographically targeted population (GNM area) over a short period of time and to evaluate the role of households in the transmission of SARS-CoV-2.

This measurement, based on a random sample, could make it possible to consolidate estimates obtained from molecular biology data (qRT-PCR) or the number of hospitalizations and/or deaths.

In addition, in vitro neutralization tests will allow an initial assessment of the ability of the detected antibodies to protect against SARS-CoV-2.

Combined with other similar studies (COVAL Paris, Epicov, ...) it will make it possible to measure the heterogeneity of virus penetration at the national level and to consolidate symptom association profiles.

All of the results (detection of cases of infection, particularly those that have not experienced symptoms, estimation of the number of people protected against a new infection (neutralisation results)) will in turn feed into mathematical models of the SEIR type (Susceptible, Exposed, Infected, Recovered).

ELIGIBILITY:
Inclusion Criteria:

* Person who has received full information about the research organization and signed informed consent
* Person residing in the Grand Nancy Metropolitan area
* Person aged at least 5 years on 1 June 2020 and weighing more than 7 kg

Exclusion Criteria:

* Children under 5 years of age at the time of collection
* Person referred to in Articles L1121-8 of the Public Health Code. A person of full age who is subject to a legal protection measure (guardianship, curatorship, legal protection).

Adult person unable to give consent

- Persons deprived of their liberty by a judicial or administrative decision, persons under psychiatric care pursuant to articles L. 3212-1 and L. 3213-1.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2006 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Anti-SARS-CoV-2 IgT (IgM/IgA/IgG) seropositivity | through study completion, an average of 4 hours
  Anti-SARS-CoV-2 IgT seropositivity of the individuals tested in the population of the Grand Nancy Metropolitan area

SECONDARY OUTCOMES:
Proportion of asymptomatic, symptomatic cases among seropositive people | through study completion, an average of 4 hours
  To estimate the proportion of occurrence of an episode of clinical symptoms since the beginning of the epidemic among seropositive people using self report questionnaires.
Proportion of asymptomatic cases among seropositive people | through study completion, an average of 4 hours
  To estimate the proportion of asymptomatic cases (asymptomatic fraction) by the proportion of seropositive individuals who did not show any sign or symptom of COVID-19 since the beginning of the epidemic in France (mid-February).
Identification of risk groups - Anti-SARS-CoV-2 IgT seropositivity by age, sex and as a function of weight status, smoking status, work activity and social status. | through study completion, an average of 4 hours
  To understand susceptibility factors to infection by comparing infected and uninfected persons on the basis of age, sex, weight status, smoking status, occupation and education.
Proportion of seropositive subjects according to the level of social disadvantage measured by the EPICES score | through study completion, an average of 4 hours
  Determining the prevalence of seropositive people according to the level of social disadvantage
Proportion of infected households | through study completion, an average of 4 hours
  To estimate the prevalence of infected households
Anti-SARS-CoV-2 IgT seropositivity in the household | through study completion, an average of 4 hours
  To provide knowledge on intra-household dissemination
Clinical expression patterns of infection by symptom/antibody association | through study completion, an average of 4 hours
  To develop symptom association profiles in seropositive subjects
Serological Response to Infection | through study completion, an average of 4 hours
  To study the serum distribution of seropositive people, particularly in each symptom typology group.
Anti-SARS-CoV-2 IgT seropositivity | through study completion, an average of 4 hours
  To use the results of the SARS-CoV-2 seroprevalence testing campaign and questionnaires to refine our knowledge of the current and future situation and make better projections with better calibrated mathematical models of SIR infectious diseases.
• Evaluation of serum neutralisation of persons positive for anti-SARS-CoV-2 antibodies, of the infectivity of viral strains in cell culture: percentage neutralisation compared to a viral strain not exposed to seropositive serum. | through study completion, an average of 4 hours
  10. To evaluate the in vitro neutralisation capacity of the viral infectivity of the antibodies detected.

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne Schvoerer, Principal Investigator — CHRU Nancy
Locations (1):
- Chru Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Yes